CLINICAL TRIAL: NCT05012228
Title: Molecular Mechanisms of Fibrillin/LTBP Superfamily in Renal Fibrosis and Cardiorenal
Brief Title: Molecular Mechanisms of Fibrillin/LTBP Superfamily in Renal Fibrosis and Cardiorenal Syndrome
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202101074RINC
Record Dates: First submitted 2021-08-03; First posted 2021-08-19 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Renal Fibrosis, CKD
Keywords: LTBP4

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is to understand the LTBP4 expression in human renal fibrotic tissues. The investigators will exam major location of LTBP4 expression and check any similar or discrepancy in renal fibrosis with different etiologies.

DETAILED DESCRIPTION:
The investigators will obtain the residual renal tissues with different etiologies and check the expression of LTBP4. The location and quantitation of LTBP4 in renal tissues will be checked. It will be great to understand the association between the severity of fibrosis and the expression of LTBP4 and other matrix proteins.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal kidney function, proteinuria, hematuria

Exclusion Criteria:

* N/A

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic kidney disease, which has remaining specimens in NTUH. The investigators want to use 2008-2016 specimens in Department of Pathology, NTUH.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Expression of LTBP4 in human renal fibrotic tissue | 5 years
Expression of biomarkers in human renal fibrotic tissue | 5 years
  Potential markers: eg. ROS-related proteins (8-oxodG, 4-HNE)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided